CLINICAL TRIAL: NCT02634489
Title: An Open-label, Parallel Group, Randomized, Two-way Crossover, Multiple Dose Study to Compare the Pharmacokinetic Profiles of Solifenacin Succinate and Tamsulosin HCl Following Co-administration of Single Entity Tablets and Administration of Three Different Dose Strengths of the Combination Tablet EC905
Brief Title: EC905 Pharmacokinetic Profile Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 905-CL-071; 2007-005155-41 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Phase 1; Healthy; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Bladder outlet obstruction; Overactive bladder; Urinary incontinence; Omnic OCAS®; Vesicare®; Tamsulosin hydrochloride; Solifenacin succinate
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction; Urinary Bladder, Overactive; Urinary Incontinence | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin HCl and Solifenacin Succinate (Active Comparator): Participants will receive daily doses of tamsulosin HCL and Solifenacin Succinate (3 dose strengths) as single tablets.
  Interventions: Drug: Tamsulosin HCl; Drug: Solifenacin Succinate
- EC905 (tamsulosin HCI and solifenacin succinate) (Active Comparator): Participants will receive a fixed combination tablet (3 dose strengths).
  Interventions: Drug: EC905

INTERVENTIONS:
Drug: Tamsulosin HCl — Oral
  Other Names: Omnic OCAS®
  Arms: Tamsulosin HCl and Solifenacin Succinate
Drug: Solifenacin Succinate — Oral
  Other Names: Vesicare®
  Arms: Tamsulosin HCl and Solifenacin Succinate
Drug: EC905 — Oral
  Other Names: Vesomni®
  Arms: EC905 (tamsulosin HCI and solifenacin succinate)

SUMMARY:
A study to compare the pharmacokinetics of tamsulosin HCl and solifenacin succinate after co-administration of single entity tablets and of the combination tablet EC905 under steady state conditions at three dose strengths.

DETAILED DESCRIPTION:
There will be 3 dose cohorts of 15 subjects each. In Period 1, subjects will be randomized to either receive multiple doses of both tamsulosin HCl and solifenacin succinate as single entity tablets, or the combination tablet EC905. The alternate treatment will be provided in Period 2. The cohorts will be balanced for period effects and first-order carry over effects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30.0 kg/m2.

Exclusion Criteria:

* Known or suspected hypersensitivity to tamsulosin HCl, solifenacin succinate, EC905 or any of the components of the formulations used.
* Any of the liver function tests above the upper limit of normal at repeated measurements.
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any other drug (excluding non-active hay fever).
* Subject is at risk of urinary retention based on medical history.
* A planned cataract surgery within 30 days after completion of the study.
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests.
* Abnormal pulse rate and/or blood pressure measurements at the pre-study visit as follows: pulse rate <40 or >90 bpm; mean systolic blood pressure >160 mmHg; mean diastolic blood pressure >100 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically).
* A marked baseline prolongation of QT/QTc interval after repeated measurements of 450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
* Use of any prescribed or OTC (over-the counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day).
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit.
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit.
* History of drinking more than 21 units of alcohol per week (1 unit = 270 cc of beer or 40 cc of spirits or 1 glass of wine) within 3 months prior to admission to the Clinical Unit.
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half-life. An exception is (partly) participation in Astellas study 905-CL-071, provided a washout of at least 12 days is considered prior to re-enrolment.
* Employee of the Astellas Group or CRO involved in the study.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of tamsulosin HCl and solifenacin succinate in plasma: AUCtau | Day 12
  AUCtau: area under the concentration - time curve (AUC) during the time interval between consecutive dosing
PK of tamsulosin HCl and solifenacin succinate in plasma: Cmax | Day 12
  Cmax: maximum concentration

SECONDARY OUTCOMES:
Safety profile assessed by adverse events, physical examination and vital signs, routine safety laboratory tests, and 12-lead ECG | Day 0 up to and including the post study visit (the PSV is scheduled between 7 to 14 days after (early) discharge on study day 13)
  Vital signs include blood pressure, pulse rate. Safety laboratory test includes urinalysis, hematology, and biochemistry. ECG: Electrocardiogram
PK profile Ctrough | Day 10, 11, 12, 13
  Ctrough: Trough concentration
PK profile PTR | Day 12
  PTR: Peak Trough Ratio
PK profile Tmax | Day 12
  Tmax: Time to attain Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Director Medical Sciences, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site NL1, Zuidlaren, Drenthe, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided